CLINICAL TRIAL: NCT02170610
Title: Bioavailability of BIBR 953 ZW After 150 mg of BIBR 1048 (Oral Pro-drug of BIBR 953) Administered as Capsule With and Without Coadministration of Pantoprazole as Well as Under the Influence of Food in Healthy Subjects. A Threeway Crossover, Randomised, Open Trial.
Brief Title: Bioavailability of BIBR 1048 MS With and Without Pantoprazole Under Influence of Food in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1160.34
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Pantoprazole

ARMS (3):
- BIBR 1048 MS capsule (Experimental)
  Interventions: Drug: BIBR 1048 MS
- BIBR 1048 capsule with pantoprazole (Experimental)
  Interventions: Drug: BIBR 1048 MS; Drug: Pantoprazole
- BIBR 1048 capsule with food (Experimental)
  Interventions: Drug: BIBR 1048 MS

INTERVENTIONS:
Drug: BIBR 1048 MS
Drug: Pantoprazole
  Arms: BIBR 1048 capsule with pantoprazole

SUMMARY:
To assess the extent of absorption of 150 mg of BIBR 1048 administered as capsule formulation with and without coadministration of 40 mg Pantoprazole and to assess the effect of food on rate and extent of absorption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP and local legislation
* Age ≥ 18 and ≤ 55 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding at the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History of or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of relevant orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of:

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2002-03; Primary Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under curve of BIBR 953 ZW in plasma over the time interval from 0 extrapolated to infinity) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
AUC0-tf (area under the plasma concentration-time curve of BIBR 953 ZW over the time interval from 0 to the last quantifiable data point) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
Cmax (maximum concentration of drug in plasma) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
tmax (time from dosing to when the plasma concentration reaches Cmax after extravascular doses) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug

SECONDARY OUTCOMES:
t½ (terminal elimination half life) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
MRTtot (mean time of residence of drug molecules in the body after oral dosing) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
CLtot/F (total clearance after oral administration) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug
Vz/F (Apparent volume of distribution during the terminal phase) of BIBR 953 ZW | Before and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48 and 72 hours after administration of study drug